CLINICAL TRIAL: NCT02052895
Title: Utility of Presepsin in Distinguishing Between Sepsis and SIRS (Systemic Inflammatory Response Syndrome): an Exploratory, Prospective Observational Study in Critically Ill Patients
Brief Title: Utility of Presepsin in Distinguishing Between Sepsis and SIRS
Status: Completed | Type: Observational
Sponsor: Mochida Pharmaceutical Company, Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: IVD2001
Record Dates: First submitted 2014-01-30; First posted 2014-02-03 (Estimated); Results first posted 2016-09-27 (Estimated); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: SIRS; Sepsis
Keywords: Presepsin; Sepsis; SIRS
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood plasma Blood serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Sepsis/SIRS: Patients with sepsis or SIRS
- Control: Patients without SIRS, sepsis, or end stage renal disease
- End Stage Renal Disease: Patients with end stage renal disease, without SIRS or sepsis

SUMMARY:
This is an observational study to evaluate the diagnostic accuracy of presepsin levels to discriminate between sepsis and SIRS upon presentation with critical illness compatible with either sepsis or systemic inflammatory response syndrome (SIRS).

ELIGIBILITY:
Sepsis/SIRS Patients

Inclusion Criteria:

* Male or female aged ≥ 21 years
* Appropriate clinical data to enable classification into sepsis or SIRS
* Written informed consent by the patient or legally authorized representative
* Critical illness consistent with SIRS or sepsis, to be enrolled within 18 hours of presentation

Exclusion Criteria:

* No informed consent
* Unacceptable risk imposed by extra blood sampling, such as by gross hemorrhage with a hematocrit < 20%

Control

Inclusion Criteria:

* Male or female aged ≥ 21 years
* Does not meet clinical criteria for sepsis or SIRS
* Written informed consent by the patient or legally authorized representative

Exclusion Criteria:

* No informed consent
* Unacceptable risk imposed by extra blood sampling, such as by gross hemorrhage with a hematocrit < 20%

End Stage Renal Disease

Inclusion Criteria:

* Male or female aged ≥ 21 years
* Documented diagnosis of end stage renal disease currently undergoing dialysis
* Does not meet clinical criteria for sepsis or SIRS
* Written informed consent by the patient or legally authorized representative

Exclusion Criteria:

* No informed consent
* Unacceptable risk imposed by extra blood sampling, such as by gross hemorrhage with a hematocrit < 20%

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with presentation to ICU with critical illness compatible with either sepsis or systemic inflammatory response syndrome (SIRS).
Sampling Method: Non-Probability Sample
Enrollment: 226 (Actual)
Dates: Start 2014-01; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanley Nasraway, MD, FCCM, Principal Investigator — Tufts Medical Center
Locations (2):
- United States (2):
  - Lahey Clinic, Boston, Massachusetts
  - Tufts Medical Center, Boston, Massachusetts

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sepsis/SIRS | Control | End Stage Renal Disease
Started | 196 | 15 | 15
Completed | 196 | 15 | 15
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Subjects who didn't meet inclusion/exclusion criteria were excluded.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sepsis/SIRS | Control | End Stage Renal Disease | Total
Number analyzed (Participants) | 190 | 15 | 15 | 220
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.80 (15.99) | 65.80 (13.11) | 53.70 (19.5) | 59.00 (16.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 6 | 9 | 88
  Male | 117 | 9 | 6 | 132

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Receiver Operating Characteristic Curve (ROC-AUC) of the Plasma Presepsin Concentration for Discriminating Between SIRS and Sepsis
Description: For the analysis, plasma presepsin levels on Day 0 were used and Sepsis/SIRS adjudication was made on Day 7 or day of discharge. ROC-AUC of presepsin for discriminating between SIRS and sepsis is compared to that of procalcitonin.
Time Frame: Up to 7 days
Population: Out of 196 Sepsis/SIRS patients, 6 were excluded due to inclusion/exclusion criteria violation and 4 were excluded due to insufficient data for Sepsis/SIRS adjudication
Measure: Least Squares Mean (95% Confidence Interval); unit: probability
Groups:
- Presepsin: ROC-AUC of presepsin for discriminating between Sepsis and SIRS
- Procalcitonin: ROC-AUC of procalcitonin for discriminating between Sepsis and SIRS
Arm/Group | Presepsin | Procalcitonin
Number analyzed (Participants) | 186 | 186
probability | 0.7218 [0.6455 to 0.7981] | 0.6901 [0.6130 to 0.7672]
Statistical Analysis 1: Comparison: Presepsin vs Procalcitonin; Test type: Superiority or Other; p = 0.3924, Regression, Logistic; Difference of ROC-AUC = 0.0317, 95% CI 2-sided [-0.0409 to 0.1043]

ADVERSE EVENTS:
Description: Six subjects who didn't meet inclusion/exclusion criteria were not assessed for adverse events.
Arm/Group | Sepsis/SIRS | Control | End Stage Renal Disease
Serious Adverse Events (participants affected / at risk) | 26/190 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/190 | 0/15 | 0/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sepsis/SIRS (N=190) | Control (N=15) | End Stage Renal Disease (N=15)
death (General disorders) | 26 (26) | 0 (0) | 0 (0)
Gastrointestinal hemmorage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hemorrhage (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 50 days from the time submitted to the sponsor for review. Only if the disclosure becomes an obstacle to the sponsor's business or registration or maintenance of the sponsor's invention, the sponsor may require changes to the communication and may extend the embargo.